CLINICAL TRIAL: NCT06443528
Title: Comparison of Lung Ultrasound Scores With Clinical Models for Predicting Bronchopulmonary Dysplasia：A Multi-center Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: jddyyy
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-03

CONDITIONS: Lung Ultrasound; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants with GA <32 weeks
  Interventions: Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: lung ultrasound — All enrolled infants underwent LUS examination performed by two ultrasound physicians. Monitoring included a complete lung scan in the first 24 hours of life (T0) and at day 3 (T1). All neonates underwent weekly ultrasound examinations until 36 weeks postmenstrual age (T2, T3…), so that the T2 scan was carried out at the end of the first week of life. LUS was performed according to a standardized protocol [13] when the neonate was in a quiet state, during routine clinical care to minimise discomfort. All ultrasound images and videos were digitally recorded, anonymised, and reviewed by a senior independent ultrasonographer blinded to patients' clinical information. Each lung was divided into three regions according to the anterior and posterior axillary lines and the mammary line. The regions were the upper-anterior, lower-anterior, and latera regions.

SUMMARY:
This study aimed to fill this knowledge gap and designed a multicentre cohort study to verify the hypothesis that LUS has good reliability to predict BPD in China and to compare the predictive value of LUS and clinical models for the development of BPD at different time points in infants born before and after 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants with GA <32 weeks.
2. Infants with enrollment within 24 hours from birth
3. Parental written consent is obtained.

Exclusion Criteria:

1. Complex congenital malformations or chromosomal abnormalities
2. Congenital lung diseases or congenital heart defects
3. Infants with enrollment after 24 hours from birth

Ages: 0 Weeks to 32 Weeks | Sex: All
Age Groups: Child
Study Population: Infants who meet all of the inclusion and exclusion criteria will be included
Sampling Method: Probability Sample
Enrollment: 1620 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
bronchopulmonary dysplasia | 2024.06.01-2027.06.30
  The outcome was bronchopulmonary dysplasia, as defined by the NIH in 2001 and Jensen in 2019：（1）no BPD as not receiving supplemental oxygen (O2) for 28 days or at 36 weeks;mild BPD as receiving O2 for greater than or equal to 28 days but not at 36 weeks; moderate BPD as receiving O2 for greater than or equal to28 days plus treatment with less than 30% O2 at 36 weeks; and severe BPD as receiving O2 for greater than or equal to 28 days plus greater than or equal to 30% O2 or positive pressure at 36 weeks；（2）No BPD was defined as breathing in room air at 36 weeks' PMA; grade 1 BPD as receipt of nasal cannula ≤2L/min (or hood O2); grade 2 BPD as nasal cannula >2L/min, nasal continuous positive airway pressure (CPAP), or nasal intermittent positive pressure ventilation;and grade 3 BPD as invasive mechanical ventilation

IPD SHARING:
Plan to Share IPD: No